CLINICAL TRIAL: NCT05839821
Title: Effects and Neural Mechanisms of Rhythmic Auditory Stimulation on Upper-limb Movements in Patients With Parkinson's Disease
Brief Title: Rhythmic Auditory Stimulation on Neural Activity During Finger-tapping in PD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, FAN Wei, PhD Candidate, The Hong Kong Polytechnic University
Other Study IDs: HongKongPU21037721r_20230220
Record Dates: First submitted 2023-02-24; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Acoustic Stimulation; Parkinson Disease; Electroencephalography
Keywords: Acoustic Stimulation; Parkinson Disease; Movement; Electroencephalography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD patients: Patients with Parkinson's disease
  Interventions: Behavioral: noF-noRAS; Behavioral: F-noRAS; Behavioral: noF-100RAS; Behavioral: F-100RAS; Behavioral: F-105RAS; Behavioral: F-110RAS
- Healthy controls: Healthy older adults
  Interventions: Behavioral: noF-noRAS; Behavioral: F-noRAS; Behavioral: noF-100RAS; Behavioral: F-100RAS; Behavioral: F-105RAS; Behavioral: F-110RAS

INTERVENTIONS:
Behavioral: noF-noRAS — resting state, that is, without finger-tapping and without listening to RAS
Behavioral: F-noRAS — finger-tapping without listening to RAS
Behavioral: noF-100RAS — listening to RAS with the 100% of the baseline tempo and without finger-tapping
Behavioral: F-100RAS — finger-tapping and listening to RAS with 100 % of baseline tempo
Behavioral: F-105RAS — finger-tapping and listening to RAS with 105 % of baseline tempo
Behavioral: F-110RAS — finger-tapping and listening to RAS with 110 % of baseline tempo

SUMMARY:
Introduction Bradykinesia (i.e., slow movements) is one of the most prominent symptoms of Parkinson's disease (PD) and has a negative impact on quality of life. Rhythmic auditory stimulation (RAS), a widely used and promising treatment technique, has been shown to effectively improve gait speed in PD patients. However, only few studies have explored effects and neural mechanisms of RAS on upper-limb movements. The investigators will conduct two studies to investigate effects and mechanisms of RAS on upper-limb movements in PD patients. The purpose of this study is to examine real-time neural activity when patients with PD and healthy controls listen to RAS and execute finger-tapping task simultaneously.

Methods and analysis This study will recruit patients with PD and healthy controls. Electroencephalography (EEG) will be used under six conditions related to a finger-tapping task. Two-way repeated measures analysis of variance will be performed to investigate the group and condition effects on neural mechanisms.

Study significance This study will offer evidence on RAS effects and mechanisms by investigating the changes in upper-limb movements and neural mechanisms during auditory-motor entrainment. Results from this study will provide a solid foundation for further research and clinical applications of RAS.

ELIGIBILITY:
Inclusion Criteria:

* (a) idiopathic PD diagnosed by a neurologist based on the Movement Disorders Society clinical diagnostic criteria;
* (b) the Hoehn and Yahr stage is 2 or 3, meaning that bilateral movement problems or combination with mild postural instability;
* (c) a score of Montreal Cognitive Assessment (MoCA) is equal to or higher than 21 to ensure that they understand experimental instructions;
* (d) a score of Edinburgh Handedness Inventory is above 60 to ensure that they are right-handed;
* (e) types and doses of medications remain unchanged in the past month right before participation.
* Age- and sex-matched healthy controls who filled the criteria (c) and (d) will be recruited from communities.

Exclusion Criteria:

* the presence of medical conditions or diseases that may affect hand movements, vision, or hearing based on self-report.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The spectral power analysis of Electroencephalography (EEG) | EEG will be continuously recorded during the whole experiment, which is about 20 minutes.
  The spectral power analysis (unit: watt) will be conducted
The functional connectivity analysis of Electroencephalography (EEG) | EEG will be continuously recorded during the whole experiment, which is about 20 minutes.
  The functional connectivity analysis (unit: coherence) will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Wei FAN (PhD student), MSc, Principal Investigator — Rehabilitation Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan W, Li J, Wei W, Xiao SH, Liao ZJ, Wang SM, Fong KNK. Effects of rhythmic auditory stimulation on upper-limb movements in patients with Parkinson's disease. Parkinsonism Relat Disord. 2022 Aug;101:27-30. doi: 10.1016/j.parkreldis.2022.06.020. Epub 2022 Jun 23. PMID 35763906
- [Background] Wang SM, Chan ST, Wong YL, Hsu HM, Lee CY, Check CY, Leung CK. Rhythmic auditory stimulation incorporated in training improved movements in individuals with psychotic-like experiences. Eur Arch Psychiatry Clin Neurosci. 2023 Jun;273(4):995-1005. doi: 10.1007/s00406-022-01524-3. Epub 2022 Nov 24. PMID 36422679
- [Background] Leuk JSP, Low LLN, Teo WP. An Overview of Acoustic-Based Interventions to Improve Motor Symptoms in Parkinson's Disease. Front Aging Neurosci. 2020 Aug 14;12:243. doi: 10.3389/fnagi.2020.00243. eCollection 2020. PMID 32922283
- [Background] Thaut MH, McIntosh GC, Rice RR, Miller RA, Rathbun J, Brault JM. Rhythmic auditory stimulation in gait training for Parkinson's disease patients. Mov Disord. 1996 Mar;11(2):193-200. doi: 10.1002/mds.870110213. PMID 8684391
- [Background] Koshimori Y, Thaut MH. Future perspectives on neural mechanisms underlying rhythm and music based neurorehabilitation in Parkinson's disease. Ageing Res Rev. 2018 Nov;47:133-139. doi: 10.1016/j.arr.2018.07.001. Epub 2018 Jul 10. PMID 30005957
- [Background] Dong VA, Fong KN, Chen YF, Tseng SS, Wong LM. 'Remind-to-move' treatment versus constraint-induced movement therapy for children with hemiplegic cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2017 Feb;59(2):160-167. doi: 10.1111/dmcn.13216. Epub 2016 Aug 9. PMID 27503605